CLINICAL TRIAL: NCT05485467
Title: The Role of CD34 + Stem Cells and Biological Markers of Angiogenesis in the Development of Coronary Allograft Vasculopathy in Patients After Heart Transplantation
Brief Title: The Role of CD34 + Stem Cells and Biomarkers in the Development of CAV in HTX Patients
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Gregor Poglajen, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 02
Record Dates: First submitted 2022-06-23; First posted 2022-08-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Vasculopathy; Heart Transplant Failure
Keywords: coronary allograft vasculopathy; CD34+ stem cells
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart transplant recipients: All patients will undergo coronary CT angiography and the presence of CAV will be defined in accordance with the ISHLT criteria. At the time of CT angiography, the patient will undergo a detailed clinical evaluation, and cardiac echo and we will also collect blood samples, perform extensive biochemical analysis and measure CD34+ cell count in peripheral venous blood
  Interventions: Diagnostic Test: coronary CT angiography

INTERVENTIONS:
Diagnostic Test: coronary CT angiography — Coronary CT angiography will be performed on multislice Siemens Somat Force CT scanner

SUMMARY:
Coronary allograft vasculopathy represents one of the major limiting factors of long-term survival in heart transplant recipients. While extensively researched, the underlying mechanisms of coronary allograft vasculopathy (CAV) after heart transplantation remain incompletely understood. As CD34+ cells represent one of the key determinants of coronary vascular homeostasis we investigated the potential association between CAV and CD34+ cell count in heart transplant recipients.

DETAILED DESCRIPTION:
In a single-center prospective pilot cohort study, we aim to enroll 55 adult heart transplant recipients. All patients will undergo coronary CT angiography and the presence of CAV will be defined in accordance with the ISHLT criteria. At the time of CT angiography, patient will undergo detailed clinical evaluation, cardiac echo and we will also collect blood samples, perform extensive biochemical analysis and measure CD34+ cell count in peripheral venous blood using Beckman-Coulter Navios EX flow cytometry with standard antibodies according to ISAGE protocol. Biomarkers of angiogenesis will be evaluated using Luminex assay kit.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant recipient
* age > 18 years
* signed informed consent

Exclusion Criteria:

* multiorgan transplantation
* eGFR < 30 ml/min
* known hypersensitivity to the contrast media
* history of any malignancy treated with radiation or chemotherapy
* therapy with mTOR inhibitors
* rejection > 1R within 90 days before enrollment
* G-CSF therapy within 30 days of enrollment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after heart transplantation, treated at Advanced Heart Failure and Transplantation Center, University Medical Center Ljubljana, Slovenia
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
CD34+ peripheral cell count in heart transplant recipients with and without coronary allograft vasculopathy | at the time of enrollment
  CD34+ peripheral cell count in heart transplant recipients with and without coronary allograft vasculopathy

SECONDARY OUTCOMES:
The serum levels of biomarkers of angiogenesis in heart transplant recipients with and without coronary allograft vasculopathy | at the time of enrollment
  The serum levels of biomarkers of angiogenesis (HIF 1a, SDF-1, IL-1, IL-6, TNFa, VEGF, FGF, EGF, Angiopoetin-2) in heart transplant recipients with and without coronary allograft vasculopathy

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Poglajen, MD, PhD, Principal Investigator — Advanced Heart Failure and Transplantation Center, Dept. of Cardiology, University Medical Center Ljubljana, Slovenia; Bojan Vrtovec, MD, PhD, Study Chair — bojan.vrtovec@kclj.si
Locations (1):
- Advanced Heart Failure and Transplantation Center, University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No